CLINICAL TRIAL: NCT06929728
Title: Copmaring Automatic Blood Preesure Measurments To Conventional Office Readings For Monitoring Hypertensive Patients And Predicting Hypertention Mediated Organ Damage
Brief Title: Automatic and Conventional Methods of Hypertensive Patients Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, vereena karam william hanna, Resident Doctor, Assiut University
Other Study IDs: Hypertension close monitoring
Record Dates: First submitted 2025-03-25; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Primary Hypertension
Keywords: HTN , HMOD ,BP , LVH ,LAE
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: this group use office conventional methods of blood pressure measurments 3 separate readings at different visits
  Interventions: Device: blood pressure measurments devices
- group 2: divided into 2 groups
  1. st group used home methods twice daily in morning and in evening using cuff digital machine
  2. nd group use unattended automatic office blood pressure measurments in 3 readings
  Interventions: Device: blood pressure measurments devices

INTERVENTIONS:
Device: blood pressure measurments devices — measure arterial blood pressure by arm cuff devises

SUMMARY:
comparing automatic blood pressure measurments methods with conventional office methods in follow up and monitoring of hypertensive patients and predicting hypertension mediated organ damage .

DETAILED DESCRIPTION:
Close monitoring of hypertensive patients using home and ambulatory blood pressure measurments and its role in predicting hypertention mediated organ damage. Echocardiography assessment for hypertensive patients and its important role in early detection and prevention of changes such as left ventricular hypertrophy,left atrial enlargement ,systolic and diastolic dysfunction and left ventricular mass . Microalbumiuria and early detection of renal impairment. Important role of close monitoring in management and control of hypertention and reduction of hypertensive emergencies and improvement of outcomes ,addherence to treatment , reduce of office consultation , improvement of psycosochial life ,reduce hospitalization cost and mortality rates . Digital apps has a good role in improve healthy life style and rapid detection of blood presssure changes during daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were screening for suspected hypertention or white coat hypertention .
* medically underserved population .
* primary arterial hypertention .
* high risk hypertensive patients [resistant hypertension ,patients with poor medication adherance ]

Exclusion Criteria:

* patients with secondary causes of hypertention
* patients with other cardiac diseases [heart faliure ,valvular heart diseases ]
* chronic illness affect blood pressure as chronic kideny disease .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A calculated minimum sample of 620 male and female hypertensive patients aged more than 18 years old recruited from outpatient clinic of assiut cardiology departement will be randomly assigned 1:1 design.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
predictive accuracy of automatic blood pressure measurments versus conventional office based measurments in identifying patient at risk of hypertension mediated organ damage [HMOD] . | over 6 months follow up period
  this outcomes will be assessed by measuring systolic and diastolic blood pressure using both automated devices [eg omron HEM -907] and conventional manual sphygmomanometers in a seated postion ,after 5 minutes of rest .measurments will be taken in duplicate on two separate visits ,one week apart and the average readings will be used for analysis .the presence of HMOD will be evaluated through echocardiographic assessment of left ventricular hypertrophy [LVH ] and microalbuminuria .correlation and predictive value [ sensitivity , specificity] will be calculated to compare both methods